CLINICAL TRIAL: NCT04720365
Title: Medico-economic Evaluation Rehabilitation by Serious Games at Home for the Management of Patients With Parkinson's Disease Suffering From Gait and Balance Disorders
Acronym: PARKGAME_ECO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019/0238/HP
Record Dates: First submitted 2020-12-29; First posted 2021-01-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Patients With Parkinson's Disease

STUDY DESIGN:
Intervention Model Description: Experimental, prospective, controlled, open randomized, multicenter, national research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- play-based rehabilitation (Experimental): Patients randomized in the "play-based rehabilitation" group will perform 2 to 3 gambling rehabilitation sessions at home using the Kinect® system linked to the Curapy.com platform for 12 months.
  Interventions: Device: play-based rehabilitaion
- routine care (No Intervention): Patients randomized in the "usual care" group will have their usual rehabilitation care provided by their physiotherapist.

INTERVENTIONS:
Device: play-based rehabilitaion — usual re-education treatment by their physiotherapist
  Other Names: Routine care
  Arms: play-based rehabilitation

SUMMARY:
This is a multi-center, randomized, open-label, multi-center, randomized controlled study of 80 Parkinson's disease patients with gait and balance disorders in which 40 patients will be treated with serious games, in addition to their usual care, for 12 months and 40 patients will be treated with their usual care during this period. This study will be conducted in 4 centers, all of which are expert in the management of these patients.

After randomization, each patient in the "Intervention-Rehabilitation through Toap Run" group will have to complete 2 to 3 sessions per week at home with the serious game "TOAP RUN" using the Kinect® system for 1 year.

DETAILED DESCRIPTION:
This is a multi-center, randomized, open-label, multi-center, randomized controlled study of 80 Parkinson's disease patients with gait and balance disorders in which 40 patients will be treated with serious games, in addition to their usual care, for 12 months and 40 patients will be treated with their usual care during this period. This study will be conducted in 4 centers, all of which are expert in the management of these patients.

After randomization, each patient in the "Intervention-Rehabilitation through Toap Run" group will have to complete 2 to 3 sessions per week at home with the serious game "TOAP RUN" using the Kinect® system for 1 year.

The primary endpoint is a medical-economic endpoint: the difference in incremental cost-utility ratio at 12 months between the 2 groups of patients. Costs will be assessed at inclusion, at the end of 6 and 12 months. Secondary endpoints include clinical and neurophysiological assessments, focusing on gait and balance disorders, as well as cognition and emotional state. An imaging study for patients included in the Paris-ICM center is also planned to study the effects of serious game rehabilitation on brain function.

Patients in both groups will be free to use SG at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic Parkinson's disease (according to United Kingdom Parkinson's Disease Society Brain Bank [UKPDD] criteria) ;
2. Age ≥ 18 years ;
3. Patient with gait and/or balance disorders not improved by levodopa treatment with item 12 "walking and balance" ≥ 1 of the MDS-UPDRS (Movement-Disorders Society-Unified Parkinson's disease rating scale) part II, ON levodopa and/or item 13 of "gait freezing" ≥ 1 (Goetz, Tilley et al. 2008);
4. Number of falls ≥ 2 in the previous year;
5. Stable antiparkinsonian treatments for at least 1 month prior to inclusion in the study ;
6. Patient with social health insurance ;
7. Person who voluntarily and informedly agreed to participate in the study (signed written consent) ;
8. Other medical problems that are stable or do not interfere with the proposed protocol;

Exclusion Criteria:

1. Parkinson's disease with Hoehn&Yahr stage 5 corresponding to an inability of the subject to stand or walk alone ;
2. Dementia (MMS < 24 and/or MoCA < 18) ;
3. Presence of an impulse control disorder defined by item 6 of the MDS-UPDRS part I > 2 ;
4. Absence of internet connection at home ;
5. Serious pathology interfering with the test ;
6. Estimated life expectancy of less than 2 years ;
7. Subject in a period of exclusion from further research ;
8. Persons under guardianship, curatorship or any other administrative or judicial measure of deprivation of rights and liberty ;
9. Pregnant woman or woman of childbearing age without contraceptive methods;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
The incremental cost-utility ratio at 12 months for the management of patients with Parkinson's disease using therapeutic games | at 12 months for the management of patients with Parkinson's disease using therapeutic games
  The result criterion is the additional cost in euros of a QALY gained. The QALY will be calculated from the utilities derived from the EuroQuality scale of life-5 dimensions EQ5D-3L.

SECONDARY OUTCOMES:
The frequency of falls | Through study completion, an average of 24 months
  The frequency of falls will be measured using item 12 of the Freezing of gait questionnaire (FOG-Q), with falls being absent (score=0), very rare (about 1/year, score=1), rare (about 1/ month, score=2), frequent (about 1/week, score=3) or very frequent (every day or several falls per day, score=4).
The incremental cost-effectiveness ratio of Toap Run therapeutic gambling management compared to usual management. | Through study completion, an average of 24 months
  The outcome criterion will be measured by the number of days of hospitalization at 12 and 24 months.
Cost-effectiveness ratio of falls prevention | Through study completion, an average of 24 months
  For the cost-effectiveness ratio of falls prevention, the clinical outcome criterion will be measured by the number of falls at 12 and 24 months.
Criterion for the cost-utility ratio | Through study completion, an average of 24 months
  The criterion for the cost-utility ratio at 24 months will be the QALY calculated from the utilities derived from the EuroQuality scale of life-5 dimensions EQ5D-3L.
The budgetary impact of Toap Run | Through study completion, an average of 24 months
  The budgetary impact of Toap Run in the management of Parkinson's patients will be measured by the resources directly consumed using the SNIIRAM/SNDS database (order of March 22, 2017 of the Public Health Code).
Incidence of treatment on Patients' quality of life | Through study completion, an average of 24 months
  Patients' quality of life will be assessed using the PDQ-39 scale, which is specific to Parkinson's disease.
Incidence of treatment on Motor skills | Through study completion, an average of 24 months
  Motor skills (walking and balance) will be assessed using clinically validated scales (UPDRS, Gait and Balance Scale, Freezing-of-gait questionnaire, Fear of falling)
Incidence of treatment on Neurological motor skills | Through study completion, an average of 24 months
  Neurological motor skills will be assessed using a neurophysiological evaluation (VICON® System).
Overall functioning | Through study completion, an average of 24 months
  Overall functioning will be assessed by the Global Functioning Scale (GFS).
Evaluation of usability and feasibility of SGs | Through study completion, an average of 24 months
  The usability and feasibility of SGs will be assessed through by patients' usability and feasability questionnaire.
Mood and anxiety | Through study completion, an average of 24 months
  Mood and anxiety will be assessed with the Hospital Anxiety Depression scale (HAD).
Emotional state | Through study completion, an average of 24 months
  Emotional state will be assessed with the Positive Affect Negative Affect Scale (PANAS).
The level of physical activity | Through study completion, an average of 24 months
  The level of physical activity evaluated with the International Physical Activity Questionnaire (IPAQ).
Patient and caregiver satisfaction | Through study completion, an average of 24 months
  Patient and caregiver satisfaction will be assessed through a satisfaction survey.
Physician user satisfaction | Through study completion, an average of 24 months
  Physician user satisfaction will be assessed through a satisfaction survey.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure WELTER, Professor, Principal Investigator — Rouen Uiniversity Hospital
Locations (4):
- France (4):
  - Chu Bordeaux, Bordeaux
  - Chu Lille, Lille
  - Gh Pitie Salpetriere, Paris
  - Rouen University Hospital, Rouen